CLINICAL TRIAL: NCT05509790
Title: A Phase 1 Study of LY3484356 in Chinese Patients With Estrogen Receptor Positive, HER2 Negative Locally Advanced or Metastatic Breast Cancer
Brief Title: A Study of LY3484356 in Chinese Participants With Advanced Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18291; J2J-MC-JZLF (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-08-19; First posted 2022-08-22 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Imlunestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LY3484356 Dose Level 1 (Experimental): Administered orally.
  Interventions: Drug: LY3484356
- LY3484356 Dose Level 2 (Experimental): Administered orally.
  Interventions: Drug: LY3484356

INTERVENTIONS:
Drug: LY3484356 — Administered orally.

SUMMARY:
This is a study of LY3484356 in Chinese participants with advanced breast cancer. Participants must have breast cancer that is estrogen receptor positive (ER+), HER2 negative (HER2-). The purpose of this study is to measure how much LY3484356 gets into the bloodstream and how long it takes the body to remove it. The safety and effectiveness of LY3484356 will also be studied. Participation could last up to 28 months.

ELIGIBILITY:
Inclusion Criteria:

* Native Chinese participants must be of an acceptable age to provide informed consent
* Have locally advanced (not amenable to curative treatment by surgery) or metastatic disease and be an appropriate candidate for experimental therapy in the judgment of the investigator, after available standard therapies have ceased to provide clinical benefit
* Have a diagnosis of ER+, HER2- breast cancer
* Female participants have postmenopausal status due either surgical/natural menopause or ovarian suppression
* If postmenopausal status is due to ovarian suppression, participants must have a negative serum pregnancy test and agree to use highly effective, medically approved precautions to prevent pregnancy
* Have a performance status less than or equal to (≤)1 on the Eastern Cooperative Oncology Group (ECOG) scale
* Have adequate organ function
* Must be able to swallow capsules/tablets

Exclusion Criteria:

* Have symptomatic central nervous system (CNS) metastasis and/or carcinomatous meningitis
* Have a serious concomitant systemic disorder

  * Human immunodeficiency virus (HIV) positive patients are excluded unless they are well controlled on highly active antiretroviral therapy with no evidence of autoimmune deficiency syndrome-defining opportunistic infections within the last 2 years, and cluster of differentiation 4 (CD4) count greater than (>)350 cells/microliter (μL)
  * Active hepatitis B or C virus infection
  * Severe renal impairment, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, history of major surgical resection involving the stomach or small bowel, preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in clinically significant diarrhea
* Have visceral crisis
* Have a serious cardiac condition
* Have an acute leukemia or other relevant cancers
* Females who are pregnant or lactating
* Known allergic reaction against any of the components of the study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-10-09 (Actual); Primary Completion 2024-02-18 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Plasma Concentration of LY3484356 | Time Frame: Cycle 1, Day 1 through Day 3 and Day 17 through Day 18; Cycle 2 Day 1 (Cycle 1 = 30 days, Cycle 2 = 28 days)
  PK: Plasma Concentration of LY3484356

SECONDARY OUTCOMES:
2. Percentage of Participants Who Achieve a Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR): Overall Response Rate (ORR) | Randomization to Disease Progression or Death from Any Cause (Estimated up to 28 months)
  ORR
Disease Control Rate (DCR): Percentage of Participants With a BOR of Complete Response (CR), Partial Response (PR) or Stable Disease (SD) | Randomization to Disease Progression or Death from Any Cause (Estimated up to 28 months)
  DCR
Progression-Free Survival (PFS) | Randomization to Disease Progression or Death from Any Cause (Estimated up to 28 months)
  PFS

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- China (4):
  - Wannan Medical College Yijishan Hospital, Wuhu, Anhui
  - Hunan Cancer Hospital, Changsha, Hunan
  - The Third Hospital of Nanchang, Nanchang, Jiangxi
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No